CLINICAL TRIAL: NCT01576640
Title: An Open Trial of Relapse Prevention Therapy for Smokers With Schizophrenia
Brief Title: Extended Duration Nicotine Replacement Therapy and Bupropion in Smokers With Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director, Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2008-04
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Nicotine Dependence; Schizophrenia
Keywords: Nicotine Dependence; Smoking Cessation; Relapse Prevention; Cognitive Behavioral Therapy; Schizophrenia
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Smoking Cessation | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Replapse Prevention Therapy (Other)
  Interventions: Drug: NRT; Drug: Bupropion SR 150mg bid; Other: Relapse Prevention-Oriented Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: NRT — Participants received nicotine replacement therapy in the form of nicotine gum/lozenge and nicotine patch
Drug: Bupropion SR 150mg bid — Subjects were given bupropion SR 150 mg bid throughout the course of the study.
Other: Relapse Prevention-Oriented Cognitive Behavioral Therapy — Subjects received relapse-prevention oriented cognitive behavioral therapy that was held weekly for 4 weeks, biweekly for 8 weeks, then monthly for 36 weeks.

SUMMARY:
After successfully quitting smoking, smokers with schizophrenia are vulnerable to relapse shortly after discontinuation of treatment. The purpose of this study was to assess the feasibility and effectiveness of a 12-month relapse prevention intervention in recently abstinent smokers with schizophrenia. Subjects participated in a 12-week smoking cessation phase, where they received nicotine replacement therapy, bupropion SR 150mg bid, and cognitive behavioral therapy. If, at the end of the 12 weeks, they were able to demonstrate 1 week of abstinence, they continued in the relapse prevention phase of the study, where they continued to receive nicotine replacement therapy, bupropion SR 150mg bid, and cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia or schizoaffective disorder by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria
* Reported smoking 10 or more cigarettes per day for at least the prior year
* Expressed a desire to quit smoking and a willingness to set a smoking cessation date within 4 weeks of enrollment
* Were psychiatrically stable on a fixed dose of an antipsychotic for the past 30 days or more
* Reported no active substance use disorder other than nicotine or caffeine within 6 months of enrollment

Exclusion Criteria:

* Participants with neurologic risk factors for bupropion treatment were excluded from receiving bupropion but were eligible to participate and receive short- and long-acting NRT and CBT only.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
7-Day Point Prevalence Abstinence at Month 15

SECONDARY OUTCOMES:
4-Week Continuous Abstinence at Month 15

CONTACTS AND LOCATIONS:
Locations (1):
- Schizophrenia Program of the Massachusetts General Hospital, Freedom Trail Clinic, 25 Staniford Street, Boston, Massachusetts, United States